CLINICAL TRIAL: NCT02397993
Title: Serum Lipase, Amylase and CA 19-9 Prior and After EUS-guided Fine Needle Aspiration of the Pancreas
Brief Title: Serum Parameter Prior and After EUS-guided Fine Needle Aspiration of the Pancreas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helios Albert-Schweitzer-Klinik Northeim (Other)
Responsible Party: Sponsor
Other Study IDs: Helios 6/1/15
Record Dates: First submitted 2015-03-15; First posted 2015-03-25 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Blood Specimen Collection; Biopsy, Fine-Needle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Pancreatic cells obtained by fine needle aspiration during endosonography Blood samples prior and after EUS with a assessment of CA19-9, Lipase and Amylase
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FNA, blood collection: blood collection prior to fine needle aspiration Endoscopic ultrasonography-guided fine needle aspiration of the pancreas blood collection after to fine needle aspiration
  Interventions: Procedure: blood collection; Procedure: fine needle aspiration

INTERVENTIONS:
Procedure: blood collection — blood will be taken for assessment of serum lipase, serum amylase and CA 19-9 prior to EUS-FNA
Procedure: fine needle aspiration — During endoscopic ultrasonography, fine needle aspiration will be performed for cytological analysis of the pancreas
Procedure: blood collection — blood will be taken 4h after EUS-FNA for assessment of serum lipase, serum amylase and CA 19-9

SUMMARY:
Endoscopic ultrasonography (EUS ) -guided fine needle aspiration (EUS -FNA ) of focal pancreatic lesions is an essential diagnostic procedure with high therapeutic effect in clinical routine.

The aim of this study is to determine the levels of serum lipase, serum amylase and the tumor marker CA 19-9 prior and after EUS-FNA. In animal experiments on dogs, an increase of all three parameters was observed after surgery on the pancreas. For humans, these clinically important data are not yet available .

It is assumed that the probability of pancreatitis with increased activity of lipase and amylase will rise with the number of puncture procedures as well as the size of the puncture needle. In addition, the post-interventional assessment of the tumor marker CA 19-9 could result in a false positive assumption of malignant neoplastic pancreatic lesion.

ELIGIBILITY:
Inclusion Criteria:

* independent indication for pancreatic EUS-FNA
* age ≥ 18 years
* patient able to give informed consent

Exclusion Criteria:

* Contraindications for EUS-FNA
* pregnancy
* no informed consent available
* known stenosis of esophagus or duodenum
* relevant coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with independent indication for endoscopic ultrasound-guided fine needle aspiration of the pancreas due to pancreatic disease (e.g. pancreatitis, pancreatic masses) no volunteers accepted
Sampling Method: Non-Probability Sample
Enrollment: 208 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Serum lipase | up to 24h prior to EUS-FNA and 4 hours after EUS-FNA

SECONDARY OUTCOMES:
Serum amylase | up to 24 hours prior to EUS-FNA
Serum amylase | 4 hours after EUS-FNA
CA 19-9 | up to 24 hours prior to EUS-FNA
CA 19-9 | 4 hours after EUS-FNA

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Meister, PD Dr., Principal Investigator — Helios Albert-Schweitzer-Klinik; Jan Heidemann, PD Dr., Principal Investigator — Klinikum Bielefeld; Volker Ellenrieder, Prof. Dr., Principal Investigator — University Medical Center Göttingen
Locations (3):
- Germany (3):
  - Department of Gastroenterology, University Medical Center, Göttingen, Lower Saxony
  - HELIOS Albert-Schweitzer Hospital Northeim, Northeim, Lower Saxony
  - Department of Gastroenterology, Klinikum Bielefeld, Bielefeld, North Rhine-Westphalia